CLINICAL TRIAL: NCT02801526
Title: A Randomized, Open-label, Single-dosing, 2x2 Crossover Study to Compare the Safety and Pharmacokinetics of CKD-330 (Fixed-dose Combination of Candesartan 16 mg and Amlodipine 5 mg) With Coadministration of the Two Separate Drugs in Healthy Male Volunteers (A)
Brief Title: Bioequivalence Study (Candesartan 16 mg and Amlodipine 5 mg) - A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 144BE15005
Record Dates: First submitted 2016-06-12; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan and Amlodipine (Experimental): Candesartan 16mg and Amlodipine 5mg, PO, 1days or 22days
  Interventions: Drug: Candesartan 16mg and Amlodipine 5mg
- CKD-330 (Experimental): CKD-330 16/5mg - A, PO, 1days or 22days
  Interventions: Drug: CKD-330 16/5mg - A

INTERVENTIONS:
Drug: CKD-330 16/5mg - A
  Arms: CKD-330
Drug: Candesartan 16mg and Amlodipine 5mg
  Arms: Candesartan and Amlodipine

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics of CKD-330 (fixed-dose combination of Candesartan 16 mg and Amlodipine 5 mg) with coadministration of the two separate drugs in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer in the age between 19 and 45 years old.
2. Body weight ≥ 55 kg and Body weight in the range of calculated IBW ±20%.
3. Subjects without a hereditary problems and chronic disease.
4. Subjects whose clinical laboratory test values are inside the accepted normal range.
5. Understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

1. Previous history or present of clinically significant hepatobiliary, nephrological, neurologic, respiratory, hemato-oncological, endocrine, urogenital, psychiatric, musculoskeletal, immune, otorhinolaryngological, cardiovascular system.
2. History of gastrointestinal disease or gastrointestinal surgery to affect drug absorption.
3. History of clinically significant allergies of amlodipine or candesartan or CCB or ARB or aspirin or antibiotic.
4. Subjects with galactose intolerance.
5. SBP ≥ 140 mmHg or< 90 mmHg, DBP ≥ 95 mmHg or < 60 mmHg, pulse ≥ 100 BPM.
6. AST or ALT > 2*ULN, total bilirubin > 2*ULN
7. Serum Creatinine > ULN
8. Previous history or present of drug abuse.
9. Subjects treated metabolizing enzyme inducers or inhibitors such as barbitals within 1 month prior to the first dosing.
10. Subjects treated ethical drug or herbal medicine within 2 weeks, OTC or vitamin within 1 week prior to the first dosing.
11. Subjects treated IP within 2 months prior to the first dosing.
12. Subjects with whole blood donation within 2 months or component blood donation within 1 month or blood transfusion within 1 month prior to the first dosing.
13. Alcohol > 21 units/week or cannot stop drinking.
14. Cigarette > 10 cigarettes/day.
15. Subjects with the plan dental treatment(extraction, orthodontic, nerve treatment) or any surgery(plastic surgery, eye surgery - LASIK, LASEK).
16. Not eligible to participate for the study at the discretion of investigator.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUCt | 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
  A. Candesartan: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
  B. Amlodipine: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
Cmax | 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
  A. Candesartan: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
  B. Amlodipine: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr

SECONDARY OUTCOMES:
AUCinf | 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
  A. Candesartan: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
  B. Amlodipine: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
tmax | 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
  A. Candesartan: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
  B. Amlodipine: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
t1/2β | 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
  A. Candesartan: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
  B. Amlodipine: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
CL/F | 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
  A. Candesartan: 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
  B. Amlodipine: 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, Principal Investigator — Chungnam National University Hospital